CLINICAL TRIAL: NCT01812447
Title: A Prospective, Randomized, Controlled Multicenter Clinical Study to Evaluate the Safety and Effectiveness of the Spiration® Valve System for the Single Lobe Treatment of Severe Emphysema
Brief Title: Evaluation of the Spiration® Valve System for Emphysema to Improve Lung Function
Acronym: EMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPR-03434
Record Dates: First submitted 2013-03-07; First posted 2013-03-18 (Estimated); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Emphysema
Keywords: Endobronchial Valves; Intrabronchial Valves; Bronchial Valve; Chronic Obstructive Pulmonary Disease; COPD; Pulmonary Disease, Chronic Obstructive; Bronchoscopic Lung Volume Reduction; BLVR; TLVR; Emphysema; Pulmonary Emphysema; Pathologic Process; Lung Diseases; Respiratory Tract Disease
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Pulmonary Emphysema; Pathologic Processes; Lung Diseases; Respiratory Tract Diseases | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spiration Valve System (Experimental): Subjects assigned to the treatment group will undergo a bronchoscopic procedure to have valves placed in the most diseased lobe of the lung to occlude all segments of the lobe. Subjects assigned to this group will also receive medical management.
  Interventions: Device: Spiration Valve System; Other: Medical Management
- Spiration Valve System, α-1 (Experimental): α-1 antitrypsin deficiency subjects will undergo a bronchoscopic procedure to have valves placed in the most diseased lobe of the lung to occlude all segments of the lobe. Subjects assigned to this group will also receive medical management. There is no randomization for this group.
  Interventions: Device: Spiration Valve System; Other: Medical Management
- Medical Management (Active Comparator): The control group for this study will receive medical management. This medical management group will be evaluated and followed in the same manner as the treatment group, but without having a bronchoscopic procedure.
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: Spiration Valve System — Subjects assigned to the treatment group will undergo a bronchoscopic procedure to have valves placed in the most diseased lobe of the lung to occlude all segments of the lobe.
  Arms: Spiration Valve System; Spiration Valve System, α-1
Other: Medical Management — Stable management is based on the ACP/ACCP/ATS/ERS Guidelines for Management of Stable COPD. Medical management will include management of COPD medications, oxygen use, and pulmonary rehabilitation.

SUMMARY:
EMPROVE is a multicenter, prospective, randomized, controlled study designed to evaluate the safety and long-term effectiveness of the Spiration Valve System in patients with emphysema.

Patients appropriate for the EMPROVE study are those who are currently on medical treatment but still symptomatic.

EMPROVE also accepts α-1 antitrypsin deficiency patients.

DETAILED DESCRIPTION:
The Spiration Valve is a small, one-way valve that is used to block air from entering diseased portions of the lung. This helps to reduce the volume in diseased lung due to hyperinflation. Volume reduction of diseased lung has been shown to improve lung function and other quality of life measures for people living with emphysema.

The Spiration Valve is placed in the diseased section of the lungs using a tool called a bronchoscope. A bronchoscope is a small tube that has a camera on the end. The bronchoscope enters the lungs through the mouth. The Spiration Valve is delivered and placed in the targeted airways via another thin tube called a catheter that travels through the bronchoscope.

* Once in place, the Spiration Valve expands and contracts with breathing, creating a complete seal around the airway
* The seal blocks air from entering the target lobe while at the same time allowing trapped air and fluids to escape.
* This causes the diseased (hyper-inflated) lung to reduce in volume or collapse
* Studies have shown volume reduction may allow healthier lung to function better
* More information and a description of the Spiration Valve System can be found on the EMPROVE clinical trial website, www.EmphysemaTrial.com

Safety and outcomes of the Spiration Valve System in emphysema have been published in several peer-reviewed journals. The articles listed below represent a summary of existing literature regarding the use of the Spiration Valve System for the treatment of emphysema. The selected articles are being provided to help understand the body of data describing the use of the Spiration Valve System.

1. Unilateral Versus Bilateral Endoscopic Lung Volume Reduction: A Comparative Case Study, NCT00995852

   Eberhardt R, Gompelmann D, Schuhmann M, Heussel CP, Herth FJ. Complete unilateral vs partial bilateral endoscopic lung volume reduction in patients with bilateral lung emphysema. Chest. 2012 Oct;142(4):900-908
2. Clinical Trial to Evaluate the Safety and Effectiveness of the IBV® Valve System for the Treatment of Severe Emphysema (IBV®Valve), NCT00475007

   Wood DE, Nader DA, Springmeyer SC, Elstad MR, Coxson HO, Chan A, Rai NS, Mularski RA, Cooper CB, Wise RA, Jones PW, Mehta AC, Gonzalez X, Sterman DH; IBV Valve Trial Research Team. The IBV Valve trial: a multicenter, randomized, double-blind trial of endobronchial therapy for severe emphysema. J Bronchology Interv Pulmonol. 2014 Oct;21(4):288-297
3. European Multi-Center Post Market Study of the IBV Valve System, NCT00880724

Ninane V, Geltner C, Bezzi M, Foccoli P, Gottlieb J, Welte T, Seijo L, Zulueta JJ, Munavvar M, Rosell A, Lopez M, Jones PW, Coxson HO, Springmeyer SC, Gonzalez X. Multicentre European study for the treatment of advanced emphysema with bronchial valves. Eur Respir J. 2012 Jun;39(6):1319-1325

ELIGIBILITY:
Inclusion Criteria:

* Subject has severe and heterogeneous emphysema with severe dyspnea
* Subject certified to meet the criteria of ATS/ERS guidelines for management of stable COPD
* Subject must be able to demonstrate physical ability to participate in the study by performing a 6-minute walk distance of ≥ 140 m
* Subject has abstained from cigarette smoking for 4 months and is willing to abstain throughout the study
* Pulmonary Function Testing Results (PFT's) demonstrate:

  * FEV1 ≤ 45% of predicted
  * RV ≥ 150% of predicted
  * TLC ≥ 100% of predicted

Exclusion Criteria:

* Patient has a BMI < 15 kg/m2
* Arterial Blood Gas Level (ABG) indicates:

  * PCO2 > 55 mm Hg
  * PO2 < 45 mm Hg on room air
* Subject has a diffuse emphysema pattern
* Subject has bronchitis with sputum production > 4 Tablespoons or 60 ml per day
* Subject has an active asthma (>15 mg of prednisone daily)
* Giant bulla (> 1/3 volume of lung)
* Pulmonary hypertension
* Subject with prior major lung surgery or recent hospitalization for COPD exacerbation or respiratory infections

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness endpoint will be the difference between the treatment and control groups in the mean change in forced expiratory volume in 1 second (FEV1) | Baseline and 6 Months

SECONDARY OUTCOMES:
Target lobe volume reduction as measured by QCT | Baseline and 6 Months
Hyperinflation as measured by the ratio of Residual Volume to Total Lung Capacity (RV/TLC) | Baseline and 6 Months
Health Status as measured by St. George's Respiratory Questionnaire (SGRQ) | Baseline and 6 Months
Dyspnea as measured by Modified Medical Research Council Questionnaire (mMRC) | Baseline and 6 Months
Exercise capacity as measured by Six Minute Walk Test (6MWT) | Baseline and 6 Months
FEV1 Responders, defined as those achieving at least 15% improvement from baseline | Baseline and 6 Months

OTHER OUTCOMES:
Incidence of thoracic SAEs | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (34):
- United States (32):
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - University of California San Diego, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Miami VA Healthcare System, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Louisiana State University Hospital, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Beaumont Botsford Hospital (DCRC), Farmington Hills, Michigan
  - Cooper University Hospital, Camden, New Jersey
  - Cornell NYPH, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Kaiser Permanente Northwest Medical Center, Clackamas, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Michael DeBakey VA Medical Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fletcher Allen Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Laval University, Québec, Quebec

REFERENCES:
- [Result] Criner GJ, Delage A, Voelker K, Hogarth DK, Majid A, Zgoda M, Lazarus DR, Casal R, Benzaquen SB, Holladay RC, Wellikoff A, Calero K, Rumbak MJ, Branca PR, Abu-Hijleh M, Mallea JM, Kalhan R, Sachdeva A, Kinsey CM, Lamb CR, Reed MF, Abouzgheib WB, Kaplan PV, Marrujo GX, Johnstone DW, Gasparri MG, Meade AA, Hergott CA, Reddy C, Mularski RA, Case AH, Makani SS, Shepherd RW, Chen B, Holt GE, Martel S. Improving Lung Function in Severe Heterogenous Emphysema with the Spiration Valve System (EMPROVE). A Multicenter, Open-Label Randomized Controlled Clinical Trial. Am J Respir Crit Care Med. 2019 Dec 1;200(11):1354-1362. doi: 10.1164/rccm.201902-0383OC. PMID 31365298
- [Result] Hogarth DK, Delage A, Zgoda MA, Nsiah-Dosu S, Himes D, Reed MF. Efficacy and safety of the Spiration Valve System for the treatment of severe emphysema in patients with Alpha-1 antitrypsin deficiency (EMPROVE). Respir Med. 2024 Apr;224:107565. doi: 10.1016/j.rmed.2024.107565. Epub 2024 Feb 14. PMID 38364975
- [Result] Criner GJ, Mallea JM, Abu-Hijleh M, Sachdeva A, Kalhan R, Hergott CA, Lazarus DR, Mularski RA, Calero K, Reed MF, Nsiah-Dosu S, Himes D, Kubo H, Kinsey CM, Majid A, Hogarth DK, Kaplan PV, Case AH, Makani SS, Chen TM, Delage A, Zgoda M, Shepherd RW. Sustained Clinical Benefits of Spiration Valve System in Patients with Severe Emphysema: 24-Month Follow-Up of EMPROVE. Ann Am Thorac Soc. 2024 Feb;21(2):251-260. doi: 10.1513/AnnalsATS.202306-520OC. PMID 37948704